CLINICAL TRIAL: NCT05470946
Title: Evaluation of the Diagnostic Role of Enteroscopy in Small Intestinal Diseases at Al-Rajhi University Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maiada Mohie Eldin Ibrahim, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Diagnostic role of enteroscopy
Record Dates: First submitted 2022-07-05; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Small Intestine Disease
MeSH Terms: interventions — Double-Balloon Enteroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enteroscopy (Other): Double balloon enteroscopy
  Interventions: Device: Double balloon enteroscopy

INTERVENTIONS:
Device: Double balloon enteroscopy — Double balloon enteroscopy (EN-580T, Fujifilm, Japan)

SUMMARY:
To identify the role of enteroscopy in diagnosis and treatment of small intestinal diseases.

DETAILED DESCRIPTION:
The small bowel is vital for digestion and absorption and is located between the stomach and large bowel. Because of its anatomical position, the small bowel was originally thought to be a "blind area" beyond the reach of ordinary endoscopic examination, leading to difficulty in diagnosing smallbowel disease.

Diseases that affect the intestinal wall are called enteropathies and can be associated with chronic diarrhea, which clinically presents in that group of patients as malabsorption syndrome and can be divided into:

1. Autoimmune causes: They include celiac disease, Crohn's disease, and other autoimmune enteropathies that affect one or several areas of the intestine.
2. Drugs: Of the antihypertensive, especially olmesartan, NSAIDs, immunosuppressant, such as azathioprine, methotrexate as well as the checkpoint inhibitors, such as nivolumab
3. Radiotherapy (RT): Up to 20% of the patients exposed to RT can develop intestinal damage; it typically occurs between 1 and 6 years, post-exposure, and is dose-dependent, usually presenting when the dose exceeds5000 cGy (centi-Gray).
4. Infectious causes: They include tropical sprue, SIBO, giardiasis, Whipple's disease, human immunodeficiency virus infection and associated opportunistic germs, tuberculosis, post-viral enteropathies, and lymphocytic enteritis associated with Helicobacter pylori infection.
5. Infiltrative and neoplastic disorders: They include eosinophilic enteritis, collagenous sprue, amyloidosis, T cell or B cell lymphoma associated with enteropathies, ymphoproliferative intestinal lymphoma, and some vasoactive substance-producing neuroendocrine tumors, especially gastrinomas, VIPomas, and intestinal carcinoid tumors.
6. Miscellaneous causes: They include conditions as diverse as peptic duodenitis, food allergies, malnutrition, lymphangiectasis, common variable immunodeficiency, or idiopathic sprue, which can also cause malabsorption syndrome

For detecting neoplastic and inflammatory diseases, endoscopy is a powerful tool. However, the diagnostic yield of a routine colonoscopy examination has been reported to be as low as 15%-30% even when an appropriate histopathological examination is added with multiple biopsy specimens.

Capsule endoscopy is an innovative method for diagnosing smallbowel disease. The reported positivity rate of capsule endoscopy for diagnosing smallbowel disease is approximately 45-81% with an accuracy rate of approximately 20-30%. However, biopsy is not possible using this approach, the precise lesion location cannot be determined, and endoscopic therapy is not possible, which limit its use.

Doubleballoon enteroscopy partly overcomes the deficiencies of capsule endoscopy, enabling examination of the entire small bowel while making biopsy and therapy possible as in stenosis dilation, extracting retained capsule endoscopy, and controlling bleeding.

The diagnostic rate of doubleballoon enteroscopy for smallbowel disease ranges from 82.4% to 86.8%.

Obtaining multiple biopsy samples from gastrointestinal mucosa is important for the diagnosis of microscopic colitis, amyloidosis, eosinophilic gastroenteritis, and celiac disease since an endoscopic examination is not sensitive enough to detect characteristic findings associated with these diseases.

Approximately 0.3-10% of individuals with celiac disease (CD) will develop refractory CD (RCD), which is associated with pre-malignant/malignant lesions which can affect anywhere along the length of the small intestine such as ulcerative jejunitis and enteropathy associated T cell lymphoma (EATL). Therefore, endoscopic evaluation of the entire length of the small bowel is essential.

Over 95% of the patients with eosinophilic gastroenteritis (EGE) reportedly have detectable endoscopic abnormalities such as multiple erosions with surrounding redness so the diagnosis of EGE is based on symptoms and eosinophilic infiltration of tissues, and a biopsy with a balloon endoscope is necessary to evaluate the histology of the small intestine.

ELIGIBILITY:
Inclusion Criteria:

* • All patients will undergo gastroscopy, colonoscopy, abdominal computed tomography and/or magnetic resonance imaging, or radionuclide examination without a clear diagnosis will be subjected to enteroscopy including:

  * patients with obscure digestive tract bleeding
  * patients with obscure diarrhea
  * patients with obscure abdominal pain
  * patients with obscure weight loss
  * patients with obscure intestinal obstruction • Patients with imaging suggesting small intestinal lesions

Exclusion Criteria:

* Patients who aren't eligible for anesthesia e.g.: severe cardiovascular, respiratory dysfunction or coagulopathy.
* Patients who aren't eligible for endoscopy e.g.: fulminant colitis, acute perforation and peritonitis, and impending perforation, intestinal obstruction, recent intestinal surgery.
* Patient's refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic role of enteroscopy in small intestinal diseases | 2 years
  To assess frequency of benign and malignant lesions of small intestine by histopathpathological examination of the obtained biopsy

SECONDARY OUTCOMES:
Side effects and complications of enteroscopy | 2 years
  To report the rate of any side effects and/or complications of the procedure such as perforation and to report rate of incomplete enteroscopy and its causes

REFERENCES:
- [Background] Baggus EMR, Hadjivassiliou M, Cross S, Penny H, Urwin H, Watson S, Woodward JM, Sanders DS. How to manage adult coeliac disease: perspective from the NHS England Rare Diseases Collaborative Network for Non-Responsive and Refractory Coeliac Disease. Frontline Gastroenterol. 2019 Aug 8;11(3):235-242. doi: 10.1136/flgastro-2019-101191. eCollection 2020. PMID 32419915
- [Background] Genta RM, Sonnenberg A. The yield of colonic biopsy in the evaluation of chronic unexplained diarrhea. Eur J Gastroenterol Hepatol. 2015 Aug;27(8):963-7. doi: 10.1097/MEG.0000000000000365. PMID 26114907
- [Background] Ghoshal UC, Gwee KA. Post-infectious IBS, tropical sprue and small intestinal bacterial overgrowth: the missing link. Nat Rev Gastroenterol Hepatol. 2017 Jul;14(7):435-441. doi: 10.1038/nrgastro.2017.37. Epub 2017 May 17. PMID 28513629
- [Background] ASGE Standards of Practice Committee; Gurudu SR, Bruining DH, Acosta RD, Eloubeidi MA, Faulx AL, Khashab MA, Kothari S, Lightdale JR, Muthusamy VR, Yang J, DeWitt JM. The role of endoscopy in the management of suspected small-bowel bleeding. Gastrointest Endosc. 2017 Jan;85(1):22-31. doi: 10.1016/j.gie.2016.06.013. Epub 2016 Jun 30. No abstract available. PMID 27374798
- [Background] Kamboj AK, Oxentenko AS. Clinical and Histologic Mimickers of Celiac Disease. Clin Transl Gastroenterol. 2017 Aug 17;8(8):e114. doi: 10.1038/ctg.2017.41. PMID 28817113
- [Background] Makkar R, Lopez R, Shen B. Clinical utility of retrograde terminal ileum intubation in the evaluation of chronic non-bloody diarrhea. J Dig Dis. 2013 Oct;14(10):536-42. doi: 10.1111/1751-2980.12082. PMID 23777610
- [Background] Kinoshita Y, Ariyoshi R, Fujigaki S, Tanaka K, Morikawa T, Sanuki T. Endoscopic diagnosis of chronic diarrhea. DEN Open. 2021 Sep 28;2(1):e53. doi: 10.1002/deo2.53. eCollection 2022 Apr. PMID 35310743
- [Background] Mizumoto N, Sasaki Y, Abe Y, Yagi M, Kon T, Onozato Y, Sakai T, Ito M, Umehara M, Ueno Y. Small-bowel Capsule Endoscopic Features in Patients with Eosinophilic Gastroenteritis: Three Case Reports. Intern Med. 2021 Sep 15;60(18):2961-2965. doi: 10.2169/internalmedicine.6935-20. Epub 2021 Mar 29. PMID 33776012
- [Background] Nakano M, Oka S, Tanaka S, Igawa A, Kunihara S, Ueno Y, Ito M, Chayama K. Indications for Small-bowel Capsule Endoscopy in Patients with Chronic Abdominal Pain. Intern Med. 2017;56(12):1453-1457. doi: 10.2169/internalmedicine.56.7458. Epub 2017 Jun 15. PMID 28626168
- [Background] Rowinski SA, Christensen E. Epidemiologic and therapeutic aspects of refractory coeliac disease - a systematic review. Dan Med J. 2016 Dec;63(12):A5307. PMID 27910801
- [Background] Shin JY, Park IS, Bang BW, Kim HK, Shin YW, Kwon KS. A Case of Primary Small Bowel Melanoma Diagnosed by Single-Balloon Enteroscopy. Clin Endosc. 2017 Jul;50(4):395-399. doi: 10.5946/ce.2016.153. Epub 2017 Jun 2. PMID 28783927
- [Background] Takenaka K, Ohtsuka K, Kitazume Y, Matsuoka K, Fujii T, Nagahori M, Kimura M, Fujioka T, Araki A, Watanabe M. Magnetic resonance evaluation for small bowel strictures in Crohn's disease: comparison with balloon enteroscopy. J Gastroenterol. 2017 Aug;52(8):879-888. doi: 10.1007/s00535-016-1284-z. Epub 2016 Nov 15. PMID 27848026
- [Background] Tang L, Huang LY, Cui J, Wu CR. Effect of Double-Balloon Enteroscopy on Diagnosis and Treatment of Small-Bowel Diseases. Chin Med J (Engl). 2018 Jun 5;131(11):1321-1326. doi: 10.4103/0366-6999.232802. PMID 29786046